CLINICAL TRIAL: NCT02332707
Title: A Phase II, Randomized, Open-Label Clinical Trial to Study the Efficacy and Safety of the Combination Regimen of MK-5172 and MK-3682 With Either MK-8742 or MK-8408 in Subjects With Chronic HCV GT1 and GT2 Infection
Brief Title: Efficacy and Safety of Grazoprevir (MK-5172) and Uprifosbuvir (MK-3682) With Elbasvir (MK-8742) or Ruzasvir (MK-8408) for Chronic Hepatitis C Genotype (GT)1 and GT2 Infection (MK-3682-011)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3682-011; 2014-003304-73 (EudraCT Number); MK-3682-011 (Other: Merck Protocol Number)
Record Dates: First submitted 2015-01-06; First posted 2015-01-07 (Estimated); Results first posted 2017-12-21 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — grazoprevir; uprifosbuvir; elbasvir; ruzasvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (18):
- A1: GT1 NC GZR+UPR+EBR (8 weeks) (Experimental): In Part A, HCV GT1-infected NC participants will take GZR 100 mg + UPR 300 mg + EBR 50 mg q.d. by mouth for 8 weeks.
  Interventions: Drug: Grazoprevir; Drug: Uprifosbuvir; Drug: Elbasvir
- A2: GT1 NC GZR+UPR+RZR (8 weeks) (Experimental): In Part A, HCV GT1-infected NC participants will take GZR 100 mg + UPR 300 mg + RZR 60 mg q.d. by mouth for 8 weeks.
  Interventions: Drug: Grazoprevir; Drug: Uprifosbuvir; Drug: Ruzasvir
- A3: GT2 NC GZR+UPR+EBR (8 weeks) (Experimental): In Part A, HCV GT2-infected NC participants will take GZR 100 mg + UPR 300 mg + EBR 50 mg q.d. by mouth for 8 weeks.
  Interventions: Drug: Grazoprevir; Drug: Uprifosbuvir; Drug: Elbasvir
- A4: GT2 NC GZR+UPR+RZR (8 weeks) (Experimental): In Part A, HCV GT2-infected NC participants will take GZR 100 mg + UPR 300 mg + RZR 60 mg q.d. by mouth for 8 weeks.
  Interventions: Drug: Grazoprevir; Drug: Uprifosbuvir; Drug: Ruzasvir
- A5: GT1 NC GZR+UPR+EBR (8 weeks) (Experimental): In Part A, HCV GT1-infected NC participants will take GZR 100 mg + UPR 450 mg + EBR 50 mg q.d. by mouth for 8 weeks.
  Interventions: Drug: Grazoprevir; Drug: Uprifosbuvir; Drug: Elbasvir
- A6: GT1 NC GZR+UPR+RZR (8 weeks) (Experimental): In Part A, HCV GT1-infected NC participants will take GZR 100 mg + UPR 450 mg + RZR 60 mg q.d. by mouth for 8 weeks.
  Interventions: Drug: Grazoprevir; Drug: Uprifosbuvir; Drug: Ruzasvir
- B7: GT2 NC GZR+UPR+EBR (8 weeks) (Experimental): In Part A, HCV GT2-infected NC participants will take GZR 100 mg + UPR 450 mg + EBR 50 mg q.d. by mouth for 8 weeks.
  Interventions: Drug: Grazoprevir; Drug: Uprifosbuvir; Drug: Elbasvir
- A8: GT2 NC GZR+UPR+RZR (8 weeks) (Experimental): In Part A, HCV GT2-infected NC participants will take GZR 100 mg + UPR 450 mg + RZR 60 mg q.d. by mouth for 8 weeks. In Part B, HCV GT2-infected NC participants will take 2 FDC tablets containing UPR 225 mg + GZR 50 mg + RZR 30 mg per tablet q.d. by mouth for 8 weeks.
  Interventions: Drug: Grazoprevir; Drug: Uprifosbuvir; Drug: Ruzasvir
- B9: GT1 NC GZR+UPR+RZR (12 weeks) (Experimental): In Part B, HCV GT1-infected NC participants will take 2 FDC tablets containing UPR 225 mg + GZR 50 mg + RZR 30 mg per tablet q.d. by mouth for 12 weeks.
  Interventions: Drug: Grazoprevir; Drug: Uprifosbuvir; Drug: Ruzasvir; Drug: Uprifosbuvir (+) Grazoprevir (+) Ruzasvir
- B10: GT2 NC GZR+UPR+RZR (8 weeks) + RBV (Experimental): In Part B, HCV GT2-infected NC participants will take 2 FDC tablets containing UPR 225 mg + GZR 50 mg + RZR 30 mg per tablet q.d. by mouth for 8 weeks. Participants will also take RBV b.i.d. at a total daily dose of 800-1600 mg based on body weight.
  Interventions: Drug: Grazoprevir; Drug: Uprifosbuvir; Drug: Ruzasvir; Drug: Uprifosbuvir (+) Grazoprevir (+) Ruzasvir; Drug: Ribavirin
- B11: GT2 NC GZR+UPR+RZR (12 weeks) (Experimental): In Part B, HCV GT2-infected NC participants will take 2 FDC tablets containing UPR 225 mg + GZR 50 mg + RZR 30 mg per tablet q.d. by mouth for 12 weeks.
  Interventions: Drug: Grazoprevir; Drug: Uprifosbuvir; Drug: Ruzasvir; Drug: Uprifosbuvir (+) Grazoprevir (+) Ruzasvir
- B12: GT1 C GZR+UPR+RZR (8 weeks) (Experimental): In Part B, HCV GT1-infected C participants will take 2 FDC tablets containing UPR 225 mg + GZR 50 mg + RZR 30 mg per tablet q.d. by mouth for 8 weeks.
  Interventions: Drug: Grazoprevir; Drug: Uprifosbuvir; Drug: Ruzasvir; Drug: Uprifosbuvir (+) Grazoprevir (+) Ruzasvir
- B13: GT1 C GZR+UPR+RZR (12 weeks) (Experimental): In Part B, HCV GT1-infected C participants will take 2 FDC tablets containing UPR 225 mg + GZR 50 mg + RZR 30 mg per tablet q.d. by mouth for 12 weeks.
  Interventions: Drug: Grazoprevir; Drug: Uprifosbuvir; Drug: Ruzasvir; Drug: Uprifosbuvir (+) Grazoprevir (+) Ruzasvir
- B14: GT2 C GZR+UPR+RZR (12 weeks) (Experimental): In Part B, HCV GT2-infected C participants will take 2 FDC tablets containing UPR 225 mg + GZR 50 mg + RZR 30 mg per tablet q.d. by mouth for 12 weeks.
  Interventions: Drug: Grazoprevir; Drug: Uprifosbuvir; Drug: Ruzasvir; Drug: Uprifosbuvir (+) Grazoprevir (+) Ruzasvir
- B15: GT2 C GZR+UPR+RZR (12 weeks) + RBV (Experimental): In Part B, HCV GT2-infected C participants will take 2 FDC tablets containing UPR 225 mg + GZR 50 mg + RZR 30 mg per tablet q.d. by mouth for 12 weeks. Participants will also take RBV b.i.d. at a total daily dose of 800-1600 mg based on body weight.
  Interventions: Drug: Grazoprevir; Drug: Uprifosbuvir; Drug: Ruzasvir; Drug: Uprifosbuvir (+) Grazoprevir (+) Ruzasvir; Drug: Ribavirin
- B16: GT2 C GZR+UPR+RZR (16 weeks) (Experimental): In Part B, HCV GT2-infected C participants will take 2 FDC tablets containing UPR 225 mg + GZR 50 mg + RZR 30 mg per tablet q.d. by mouth for 16 weeks.
  Interventions: Drug: Grazoprevir; Drug: Uprifosbuvir; Drug: Ruzasvir; Drug: Uprifosbuvir (+) Grazoprevir (+) Ruzasvir
- B6: GT1 NC GZR+UPR+RZR (8 weeks) (Experimental): In Part B, HCV GT1-infected NC participants will take 2 FDC tablets containing UPR 225 mg + GZR 50 mg + RZR 30 mg per tablet q.d. by mouth for 8 weeks.
  Interventions: Drug: Uprifosbuvir (+) Grazoprevir (+) Ruzasvir
- B8: GT2 NC GZR+UPR+RZR (8 weeks) (Experimental): In Part B, HCV GT2-infected NC participants will take 2 FDC tablets containing UPR 225 mg + GZR 50 mg + RZR 30 mg per tablet q.d. by mouth for 8 weeks.
  Interventions: Drug: Uprifosbuvir (+) Grazoprevir (+) Ruzasvir

INTERVENTIONS:
Drug: Grazoprevir — One GZR 100 mg tablet (Part A), or 2 FDC tablets containing GZR 50 mg per tablet (Part B), taken q.d.by mouth.
  Other Names: MK-5172
  Arms: A1: GT1 NC GZR+UPR+EBR (8 weeks); A2: GT1 NC GZR+UPR+RZR (8 weeks); A3: GT2 NC GZR+UPR+EBR (8 weeks); A4: GT2 NC GZR+UPR+RZR (8 weeks); A5: GT1 NC GZR+UPR+EBR (8 weeks); A6: GT1 NC GZR+UPR+RZR (8 weeks); A8: GT2 NC GZR+UPR+RZR (8 weeks); B10: GT2 NC GZR+UPR+RZR (8 weeks) + RBV; B11: GT2 NC GZR+UPR+RZR (12 weeks); B12: GT1 C GZR+UPR+RZR (8 weeks); B13: GT1 C GZR+UPR+RZR (12 weeks); B14: GT2 C GZR+UPR+RZR (12 weeks); B15: GT2 C GZR+UPR+RZR (12 weeks) + RBV; B16: GT2 C GZR+UPR+RZR (16 weeks); B7: GT2 NC GZR+UPR+EBR (8 weeks); B9: GT1 NC GZR+UPR+RZR (12 weeks)
Drug: Uprifosbuvir — Two or 3 UPR 150 mg (300 mg and 450 mg total daily dose) tablets (Part A), or 2 FDC tablets containing UPR 225 mg (Part B), taken q.d. by mouth.
  Other Names: MK-3682
  Arms: A1: GT1 NC GZR+UPR+EBR (8 weeks); A2: GT1 NC GZR+UPR+RZR (8 weeks); A3: GT2 NC GZR+UPR+EBR (8 weeks); A4: GT2 NC GZR+UPR+RZR (8 weeks); A5: GT1 NC GZR+UPR+EBR (8 weeks); A6: GT1 NC GZR+UPR+RZR (8 weeks); A8: GT2 NC GZR+UPR+RZR (8 weeks); B10: GT2 NC GZR+UPR+RZR (8 weeks) + RBV; B11: GT2 NC GZR+UPR+RZR (12 weeks); B12: GT1 C GZR+UPR+RZR (8 weeks); B13: GT1 C GZR+UPR+RZR (12 weeks); B14: GT2 C GZR+UPR+RZR (12 weeks); B15: GT2 C GZR+UPR+RZR (12 weeks) + RBV; B16: GT2 C GZR+UPR+RZR (16 weeks); B7: GT2 NC GZR+UPR+EBR (8 weeks); B9: GT1 NC GZR+UPR+RZR (12 weeks)
Drug: Elbasvir — One EBR 50 mg tablet (Part A), taken q.d. by mouth.
  Other Names: MK-8742
  Arms: A1: GT1 NC GZR+UPR+EBR (8 weeks); A3: GT2 NC GZR+UPR+EBR (8 weeks); A5: GT1 NC GZR+UPR+EBR (8 weeks); B7: GT2 NC GZR+UPR+EBR (8 weeks)
Drug: Ruzasvir — Six RZR 10 mg (60 mg total daily dose) capsules (Part A), or 2 FDC tablets containing RZR 30 mg per tablet (Part B), taken q.d. by mouth.
  Other Names: MK-8408
  Arms: A2: GT1 NC GZR+UPR+RZR (8 weeks); A4: GT2 NC GZR+UPR+RZR (8 weeks); A6: GT1 NC GZR+UPR+RZR (8 weeks); A8: GT2 NC GZR+UPR+RZR (8 weeks); B10: GT2 NC GZR+UPR+RZR (8 weeks) + RBV; B11: GT2 NC GZR+UPR+RZR (12 weeks); B12: GT1 C GZR+UPR+RZR (8 weeks); B13: GT1 C GZR+UPR+RZR (12 weeks); B14: GT2 C GZR+UPR+RZR (12 weeks); B15: GT2 C GZR+UPR+RZR (12 weeks) + RBV; B16: GT2 C GZR+UPR+RZR (16 weeks); B9: GT1 NC GZR+UPR+RZR (12 weeks)
Drug: Uprifosbuvir (+) Grazoprevir (+) Ruzasvir — Two FDC tablets, each containing GZR 50 mg + UPR 225 mg + RZR 30 mg (Part B), taken q.d. by mouth.
  Other Names: MK-3682B
  Arms: B10: GT2 NC GZR+UPR+RZR (8 weeks) + RBV; B11: GT2 NC GZR+UPR+RZR (12 weeks); B12: GT1 C GZR+UPR+RZR (8 weeks); B13: GT1 C GZR+UPR+RZR (12 weeks); B14: GT2 C GZR+UPR+RZR (12 weeks); B15: GT2 C GZR+UPR+RZR (12 weeks) + RBV; B16: GT2 C GZR+UPR+RZR (16 weeks); B6: GT1 NC GZR+UPR+RZR (8 weeks); B8: GT2 NC GZR+UPR+RZR (8 weeks); B9: GT1 NC GZR+UPR+RZR (12 weeks)
Drug: Ribavirin — RBV 200 mg capsules taken b.i.d. at a total daily dose of 800-1400 mg based on participant body weight.
  Other Names: Rebetol®
  Arms: B10: GT2 NC GZR+UPR+RZR (8 weeks) + RBV; B15: GT2 C GZR+UPR+RZR (12 weeks) + RBV

SUMMARY:
This is a randomized, three-part, open-label trial of grazoprevir (GZR; MK-5172) (100 mg) and uprifosbuvir (UPR; MK-3682) (300 mg or 450 mg), with either elbasvir (EBR; MK-8742) (50 mg) or ruzasvir (RZR; MK-8408) (60 mg), and with or without ribavirin (RBV), in treatment-naïve (TN) cirrhotic (C) or non-cirrhotic (NC) hepatitis C virus (HCV) participants with chronic HCV genotype (GT) 1 or GT2 infection. Part A will consist of 8 arms to evaluate the safety of dose combinations. In Part B, participants will take 2 UPR+GZR+RZR fixed dose combination (FDC) tablets once daily (q.d.) by mouth, with or without twice-daily (b.i.d.) RBV (200 mg capsules; weight-based dosing). Participants who relapse following completion of therapy in Part A will be offered the option of retreatment with 16 weeks of UPR+GZR+RZR with RBV in Part C (data obtained from Part C will not be used in the analysis of outcome measures).

DETAILED DESCRIPTION:
In Part A, study therapy will be administered as separate products, each taken q.d. by mouth. In Part B and Part C, participants will take 2 FDC tablets containing UPR 225 mg + GZR 50 mg + RZR 30 mg q.d. by mouth.

ELIGIBILITY:
Inclusion Criteria:

Parts A and B:

* Previously untreated chronic HCV GT1 or GT2 with no evidence of non-typeable or mixed genotype infection
* Has HCV ribonucleic acid (RNA) >= 10,000 IU/mL in peripheral blood at the time of screening
* Is NC (Part A and B)
* Is HCV treatment naïve (defined as no prior exposure to any interferon, ribavirin, or other approved or experimental HCV-specific direct-acting antiviral agent
* Is of non-childbearing potential or agrees to avoid becoming pregnant or impregnating a partner beginning at least 2 weeks prior to administration of the initial dose of study drug and either for 14 days after the last dose of study drug if not taking RBV or for 6 months after the last dose of study drug if taking RBV (or longer if dictated by local regulations). If not abstinent from heterosexual activity, participants in Part A must use 2 acceptable forms of barrier contraception whereas participants in Part B must use 2 acceptable forms of contraception which may include oral contraceptives

Part B only:

* Has cirrhosis of the liver
* If coinfected with human immunodeficiency virus (HIV) is not currently on antiretroviral therapy (ART) and has no plans to initiate ART treatment while participating in this study OR has well controlled HIV on ART (the ART regimen must contain only the following antiretroviral medications: tenofovir, abacavir, lamivudine, emtricitabine, raltegravir, dolutegravir, and rilpivirine with no dose modifications or changes in drugs in the 4 weeks prior to study entry [Day 1])
* Has at least one viable ART regimen alternative beyond their current regimen in the event of HIV virologic failure and the development of antiretroviral drug resistance

Exclusion Criteria:

Parts A, B, and C (unless noted otherwise):

* Has evidence of decompensated liver disease manifested by the presence of or history of ascites, esophageal or gastric variceal bleeding, hepatic encephalopathy or other signs or symptoms of advanced liver disease
* For cirrhotics (Part B only), participants who are Child-Pugh Class B or C or who have a Pugh-Turcotte (CPT) score >5
* Is coinfected with hepatitis B virus
* Is coinfected with HIV (Part A only)
* If coinfected with HIV (Part B only), has a history of opportunistic infection in the preceding 6 months prior to screening
* Has a history of malignancy <=5 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer or carcinoma in situ; or is under evaluation for other active or suspected malignancy
* Has cirrhosis and has had liver imaging within 6 months of Day 1 showing evidence of hepatocellular carcinoma (HCC) or is under evaluation for HCC
* Has clinically-relevant drug or alcohol abuse within 12 months of screening
* Pregnant or breast-feeding, or expecting to conceive or donate eggs from at least 2 weeks prior to Day 1 and 90 days after the last dose of study medication, or longer if dictated by local regulations
* Has any of the following conditions:
* organ transplants (including hematopoietic stem cell transplants) other than cornea and hair
* poor venous access that precludes routine peripheral blood sampling required for this trial
* has a history of gastric surgery (e.g., stapling, bypass) or history of malabsorption disorders (e.g., celiac sprue disease)
* current or history of any clinically significant cardiac abnormalities/dysfunction, including but not limited to: angina, congestive heart failure, myocardial infarction, pulmonary hypertension, complex congenital heart disease, cardiomyopathy, significant arrhythmia, uncontrolled hypertension, a history of use of antianginal or anti-arrhythmic agents for cardiac conditions, prolonged electrocardiogram (ECG) QTc interval (>470 ms for males or >480 ms for females by the Fridericia formula) at the screening visit, personal or family history of Torsade de pointes
* chronic pulmonary disease, including but not limited to: clinically significant chronic obstructive pulmonary disease, interstitial lung disease, pulmonary fibrosis, sarcoidosis
* central nervous system (CNS) trauma requiring intubation, intracranial pressure monitoring, brain meningeal or skull surgery, or resulting in seizure, coma, permanent neurologic deficits, abnormal brain imaging, or cerebral spinal fluid (CSF) leak. Prior brain hemorrhage and/or intracranial aneurysms (whether adequately repaired or not)
* a current, or history of, seizure disorder unless seizure was >10 years ago, a single isolated event, no history of or current use of anti-seizure medications prescribed, and a normal neurological examination is documented in trial files within 6 months of Day 1
* a history of stroke or transient ischemic attack
* a history of a medical/surgical condition that resulted in hospitalization within the 3 months prior to enrollment, other than for minor elective procedures
* a medical/surgical conditions that may result in a need for hospitalization during the period of the study
* any medical condition requiring, or likely to require, chronic systemic administration of corticosteroids, tumor necrosis factor (TNF) antagonists, or other immunosuppressant drugs during the course of the trial
* has any condition, prestudy laboratory or ECG abnormality or history of any illness, which, in the opinion of the investigator, might confound the results of the study or pose additional risk in administering the study drugs to the subject
* experiences a life-threatening serious adverse event (SAE) during the screening period
* evidence of history of chronic hepatitis not caused by HCV, including but not limited to nonalcoholic steatohepatitis (NASH), drug-induced hepatitis, hemochromatosis, Wilson's disease, α1-antitrypsin deficiency, alcoholic liver disease, and autoimmune hepatitis
* hemoglobinopathy, including, but not limited to, thalassemia major (Parts B and C only) Parts B and C only: is a male whose female partner(s) is/are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 443 (Actual)
Dates: Start 2015-01-22 (Actual); Primary Completion 2016-09-16 (Actual); Study Completion 2016-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Lawitz E, Buti M, Vierling JM, Almasio PL, Bruno S, Ruane PJ, Hassanein TI, Muellhaupt B, Pearlman B, Jancoriene L, Gao W, Huang HC, Shepherd A, Tannenbaum B, Fernsler D, Li JJ, Grandhi A, Liu H, Su FH, Wan S, Dutko FJ, Nguyen BT, Wahl J, Robertson MN, Barr E, Yeh WW, Plank RM, Butterton JR, Yoshida EM. Safety and efficacy of a fixed-dose combination regimen of grazoprevir, ruzasvir, and uprifosbuvir with or without ribavirin in participants with and without cirrhosis with chronic hepatitis C virus genotype 1, 2, or 3 infection (C-CREST-1 and C-CREST-2, part B): two randomised, phase 2, open-label trials. Lancet Gastroenterol Hepatol. 2017 Nov;2(11):814-823. doi: 10.1016/S2468-1253(17)30163-2. Epub 2017 Aug 10. PMID 28802814
- [Derived] Gane EJ, Pianko S, Roberts SK, Thompson AJ, Zeuzem S, Zuckerman E, Ben-Ari Z, Foster GR, Agarwal K, Laursen AL, Gerstoft J, Gao W, Huang HC, Fitzgerald B, Fernsler D, Li JJ, Grandhi A, Liu H, Su FH, Wan S, Zeng Z, Chen HL, Dutko FJ, Nguyen BT, Wahl J, Robertson MN, Barr E, Yeh WW, Plank RM, Butterton JR, Esteban R. Safety and efficacy of an 8-week regimen of grazoprevir plus ruzasvir plus uprifosbuvir compared with grazoprevir plus elbasvir plus uprifosbuvir in participants without cirrhosis infected with hepatitis C virus genotypes 1, 2, or 3 (C-CREST-1 and C-CREST-2, part A): two randomised, phase 2, open-label trials. Lancet Gastroenterol Hepatol. 2017 Nov;2(11):805-813. doi: 10.1016/S2468-1253(17)30159-0. Epub 2017 Aug 10. PMID 28802816

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted at 95 study sites in Asia, the European Union, and North America.
Pre-assignment Details: The "Number Started" row reflects the number of randomized participants who received study treatment. A total of 443 participants were randomized but 1 participant withdrew consent prior to receiving any study treatment.
Groups:
- A1: GT1 NC GZR+UPR+EBR (8 Weeks): In Part A, Hepatitis C virus (HCV) genotype (GT)1-infected non-cirrhotic (NC) participants took grazoprevir (GZR) 100 mg + uprifosbuvir (UPR) 300 mg + elbasvir (EBR) 50 mg once daily (q.d.) by mouth for 8 weeks.
- A2: GT1 NC GZR+UPR+RZR (8 Weeks): In Part A, HCV GT1-infected NC participants took GZR 100 mg + UPR 300 mg + ruzasvir (RZR) 60 mg q.d. by mouth for 8 weeks.
- A3: GT2 NC GZR+UPR+EBR (8 Weeks): In Part A, HCV GT2-infected NC participants took GZR 100 mg + UPR 300 mg + EBR 50 mg q.d. by mouth for 8 weeks.
- A4: GT2 NC GZR+UPR+RZR (8 Weeks): In Part A, HCV GT2-infected NC participants took GZR 100 mg + UPR 300 mg + RZR 60 mg q.d. by mouth for 8 weeks.
- A5: GT1 NC GZR+UPR+EBR (8 Weeks): In Part A, HCV GT1-infected NC participants took GZR 100 mg + UPR 450 mg + EBR 50 mg q.d. by mouth for 8 weeks.
- A6: GT1 NC GZR+UPR+RZR (8 Weeks): In Part A, HCV GT1-infected NC participants took GZR 100 mg + UPR 450 mg + RZR 60 mg q.d. by mouth for 8 weeks.
- A7: GT2 NC GZR+UPR+EBR (8 Weeks): In Part A, HCV GT2-infected NC participants took GZR 100 mg + UPR 450 mg + EBR 50 mg q.d. by mouth for 8 weeks.
- A8: GT2 NC GZR+UPR+RZR (8 Weeks): In Part A, HCV GT2-infected NC participants took GZR 100 mg + UPR 450 mg + RZR 60 mg q.d. by mouth for 8 weeks.
- B9: GT1 NC GZR+UPR+RZR (12 Weeks): In Part B, HCV GT1-infected NC participants took 2 fixed dose combination (FDC) tablets containing GZR 50 mg + UPR 225 mg + RZR 30 mg per tablet q.d. by mouth for 12 weeks.
- B10: GT2 NC GZR+UPR+RZR (8 Weeks) + RBV: In Part B, HCV GT2-infected NC participants took 2 FDC tablets containing GZR 50 mg + UPR 225 mg + RZR 30 mg per tablet q.d. by mouth for 8 weeks. Participants will also take RBV b.i.d. at a total daily dose of 800-1600 mg based on body weight.
- B11: GT2 NC GZR+UPR+RZR (12 Weeks): In Part B, HCV GT2-infected NC participants took 2 FDC tablets containing GZR 50 mg + UPR 225 mg + RZR 30 mg per tablet q.d. by mouth for 12 weeks.
- B12: GT1 C GZR+UPR+RZR (8 Weeks): In Part B, HCV GT1-infected C participants took 2 FDC tablets containing GZR 50 mg + UPR 225 mg + RZR 30 mg per tablet q.d. by mouth for 8 weeks.
- B13: GT1 C GZR+UPR+RZR (12 Weeks): In Part B, HCV GT1-infected C participants took 2 FDC tablets containing GZR 50 mg + UPR 225 mg + RZR 30 mg per tablet q.d. by mouth for 12 weeks.
- B14: GT2 C GZR+UPR+RZR (12 Weeks): In Part B, HCV GT2-infected C participants took 2 FDC tablets containing GZR 50 mg + UPR 225 mg + RZR 30 mg per tablet q.d. by mouth for 12 weeks.
- B15: GT2 C GZR+UPR+RZR (12 Weeks) + RBV: In Part B, HCV GT2-infected C participants took 2 FDC tablets containing GZR 50 mg + UPR 225 mg + RZR 30 mg per tablet q.d. by mouth for 12 weeks. Participants will also take RBV b.i.d. at a total daily dose of 800-1600 mg based on body weight.
- B16: GT2 C GZR+UPR+RZR (16 Weeks): In Part B, HCV GT2-infected C participants took 2 FDC tablets containing UPR 225 mg + GZR 50 mg + RZR 30 mg per tablet q.d. by mouth for 16 weeks.
- B6: GT1 NC GZR+UPR+RZR (8 Weeks): In Part B, HCV GT1-infected NC participants took 2 FDC tablets containing UPR 225 mg + GZR 50 mg + RZR 30 mg per tablet q.d. by mouth for 8 weeks.
- B8: GT2 NC GZR+UPR+RZR (8 Weeks): In Part B, HCV GT2-infected NC participants took 2 FDC tablets containing GZR 50 mg + UPR 225 mg + RZR 30 mg per tablet q.d. by mouth for 8 weeks.
Period: Overall Study
Arm/Group | A1: GT1 NC GZR+UPR+EBR (8 Weeks) | A2: GT1 NC GZR+UPR+RZR (8 Weeks) | A3: GT2 NC GZR+UPR+EBR (8 Weeks) | A4: GT2 NC GZR+UPR+RZR (8 Weeks) | A5: GT1 NC GZR+UPR+EBR (8 Weeks) | A6: GT1 NC GZR+UPR+RZR (8 Weeks) | A7: GT2 NC GZR+UPR+EBR (8 Weeks) | A8: GT2 NC GZR+UPR+RZR (8 Weeks) | B9: GT1 NC GZR+UPR+RZR (12 Weeks) | B10: GT2 NC GZR+UPR+RZR (8 Weeks) + RBV | B11: GT2 NC GZR+UPR+RZR (12 Weeks) | B12: GT1 C GZR+UPR+RZR (8 Weeks) | B13: GT1 C GZR+UPR+RZR (12 Weeks) | B14: GT2 C GZR+UPR+RZR (12 Weeks) | B15: GT2 C GZR+UPR+RZR (12 Weeks) + RBV | B16: GT2 C GZR+UPR+RZR (16 Weeks) | B6: GT1 NC GZR+UPR+RZR (8 Weeks) | B8: GT2 NC GZR+UPR+RZR (8 Weeks)
Started | 23 | 24 | 16 | 14 | 23 | 23 | 15 | 16 | 48 | 31 | 31 | 35 | 40 | 15 | 16 | 26 | 30 | 16
Completed | 23 | 24 | 15 | 13 | 23 | 22 | 15 | 16 | 48 | 28 | 29 | 35 | 35 | 15 | 16 | 26 | 30 | 16
Not Completed | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 2 | 0 | 5 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Baseline Population consists of all randomized participants who received study medication.
Groups:
- B9: GT1 NC GZR+UPR+RZR (12 Weeks): In Part B, HCV GT1-infected NC participants took 2 FDC tablets containing GZR 50 mg + UPR 225 mg + RZR 30 mg per tablet q.d. by mouth for 12 weeks.
- B6: GT1 NC GZR+UPR+RVR (8 Weeks): In Part B, HCV GT1-infected NC participants took 2 FDC tablets containing GZR 50 mg + UPR 225 mg + RZR 30 mg per tablet q.d. by mouth for 8 weeks.
- Total: Total of all reporting groups
Arm/Group | A1: GT1 NC GZR+UPR+EBR (8 Weeks) | A2: GT1 NC GZR+UPR+RZR (8 Weeks) | A3: GT2 NC GZR+UPR+EBR (8 Weeks) | A4: GT2 NC GZR+UPR+RZR (8 Weeks) | A5: GT1 NC GZR+UPR+EBR (8 Weeks) | A6: GT1 NC GZR+UPR+RZR (8 Weeks) | A7: GT2 NC GZR+UPR+EBR (8 Weeks) | A8: GT2 NC GZR+UPR+RZR (8 Weeks) | B9: GT1 NC GZR+UPR+RZR (12 Weeks) | B10: GT2 NC GZR+UPR+RZR (8 Weeks) + RBV | B11: GT2 NC GZR+UPR+RZR (12 Weeks) | B12: GT1 C GZR+UPR+RZR (8 Weeks) | B13: GT1 C GZR+UPR+RZR (12 Weeks) | B14: GT2 C GZR+UPR+RZR (12 Weeks) | B15: GT2 C GZR+UPR+RZR (12 Weeks) + RBV | B16: GT2 C GZR+UPR+RZR (16 Weeks) | B6: GT1 NC GZR+UPR+RVR (8 Weeks) | B8: GT2 NC GZR+UPR+RZR (8 Weeks) | Total
Number analyzed (Participants) | 23 | 24 | 16 | 14 | 23 | 23 | 15 | 16 | 48 | 31 | 31 | 35 | 40 | 15 | 16 | 26 | 30 | 16 | 442
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.2 (13.5) | 45.0 (14.5) | 49.4 (15.8) | 52.6 (11.6) | 49.0 (11.2) | 46.7 (13.9) | 52.9 (12.1) | 48.3 (8.8) | 48.8 (13.9) | 49.8 (13.0) | 55.6 (14.4) | 58.8 (9.6) | 56.9 (11.1) | 61.8 (6.8) | 59.8 (8.0) | 64.0 (9.3) | 47.4 (11.7) | 51.4 (10.8) | 52.6 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 7 | 5 | 14 | 9 | 9 | 8 | 21 | 16 | 16 | 14 | 11 | 3 | 4 | 9 | 14 | 9 | 192
  Male | 13 | 11 | 9 | 9 | 9 | 14 | 6 | 8 | 27 | 15 | 15 | 21 | 29 | 12 | 12 | 17 | 16 | 7 | 250

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Virologic Response 12 Weeks After Completing Treatment (SVR12)
Description: The percentage of participants with Hepatitis C virus (HCV) ribonucleic acid (RNA) < Lower Limit of Quantification (LLoQ) 12 weeks after completing treatment (i.e., SVR12) in each arm was determined. Plasma levels of HCV RNA levels were measured using the Roche COBAS® AmpliPrep/COBAS® TaqMan® HCV Test, v2.0 assay, which has a LLoQ of 15 IU/mL.
Time Frame: Up to 28 weeks
Population: All randomized participants who received at least 1 dose of study drug and had SVR12 results available are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- 16: GT2 C GZR+UPR+RZR (16 Weeks): In Part B, HCV GT2-infected C participants took 2 FDC tablets containing GZR 50 mg + UPR 225 mg + RZR 30 mg per tablet q.d. by mouth for 16 weeks.
Arm/Group | A1: GT1 NC GZR+UPR+EBR (8 Weeks) | A2: GT1 NC GZR+UPR+RZR (8 Weeks) | A3: GT2 NC GZR+UPR+EBR (8 Weeks) | A4: GT2 NC GZR+UPR+RZR (8 Weeks) | A5: GT1 NC GZR+UPR+EBR (8 Weeks) | A6: GT1 NC GZR+UPR+RZR (8 Weeks) | B6: GT1 NC GZR+UPR+RVR (8 Weeks) | A7: GT2 NC GZR+UPR+EBR (8 Weeks) | A8: GT2 NC GZR+UPR+RZR (8 Weeks) | B8: GT2 NC GZR+UPR+RZR (8 Weeks) | B9: GT1 NC GZR+UPR+RZR (12 Weeks) | B10: GT2 NC GZR+UPR+RZR (8 Weeks) + RBV | B11: GT2 NC GZR+UPR+RZR (12 Weeks) | B12: GT1 C GZR+UPR+RZR (8 Weeks) | B13: GT1 C GZR+UPR+RZR (12 Weeks) | B14: GT2 C GZR+UPR+RZR (12 Weeks) | B15: GT2 C GZR+UPR+RZR (12 Weeks) + RBV | 16: GT2 C GZR+UPR+RZR (16 Weeks)
Number analyzed (Participants) | 23 | 24 | 16 | 14 | 23 | 23 | 30 | 15 | 16 | 16 | 48 | 30 | 30 | 35 | 39 | 15 | 16 | 25
Percentage of Participants | 100.0 [85.2 to 100.0] | 100.0 [85.8 to 100.0] | 68.8 [41.3 to 89.0] | 71.4 [41.9 to 91.6] | 100.0 [85.2 to 100.0] | 91.3 [72.0 to 98.9] | 100.0 [88.4 to 100.0] | 60.0 [32.3 to 83.7] | 93.8 [69.8 to 99.8] | 87.5 [61.7 to 98.4] | 100.0 [92.6 to 100.0] | 83.3 [65.3 to 94.4] | 100.0 [88.4 to 100.0] | 97.1 [85.1 to 99.9] | 100.0 [91.0 to 100.0] | 100.0 [78.2 to 100.0] | 100.0 [79.4 to 100.0] | 100.0 [86.3 to 100.0]

2. Primary Outcome: Percentage of Participants Experiencing an Adverse Event (AE)
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to 18 weeks
Population: All randomized participants who received at least 1 dose of study drug are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | A1: GT1 NC GZR+UPR+EBR (8 Weeks) | A2: GT1 NC GZR+UPR+RZR (8 Weeks) | A3: GT2 NC GZR+UPR+EBR (8 Weeks) | A4: GT2 NC GZR+UPR+RZR (8 Weeks) | A5: GT1 NC GZR+UPR+EBR (8 Weeks) | A6: GT1 NC GZR+UPR+RZR (8 Weeks) | B6: GT1 NC GZR+UPR+RVR (8 Weeks) | A7: GT2 NC GZR+UPR+EBR (8 Weeks) | A8: GT2 NC GZR+UPR+RZR (8 Weeks) | B8: GT2 NC GZR+UPR+RZR (8 Weeks) | B9: GT1 NC GZR+UPR+RZR (12 Weeks) | B10: GT2 NC GZR+UPR+RZR (8 Weeks) + RBV | B11: GT2 NC GZR+UPR+RZR (12 Weeks) | B12: GT1 C GZR+UPR+RZR (8 Weeks) | B13: GT1 C GZR+UPR+RZR (12 Weeks) | B14: GT2 C GZR+UPR+RZR (12 Weeks) | B15: GT2 C GZR+UPR+RZR (12 Weeks) + RBV | 16: GT2 C GZR+UPR+RZR (16 Weeks)
Number analyzed (Participants) | 23 | 24 | 16 | 14 | 23 | 23 | 30 | 15 | 16 | 16 | 48 | 31 | 31 | 35 | 40 | 15 | 16 | 26
Percentage of Participants | 60.9 | 83.3 | 56.3 | 71.4 | 73.9 | 60.9 | 62.3 | 86.7 | 75.0 | 68.8 | 72.9 | 80.6 | 71.0 | 57.1 | 72.5 | 53.3 | 81.3 | 69.2

3. Secondary Outcome: Percentage of Participants Achieving Sustained Virologic Response 24 Weeks After Ending Study Treatment (SVR24)
Description: The percentage of participants with HCV RNA < LLoQ 24 weeks after completing treatment (i.e., SVR24) in each arm was determined. Plasma levels of HCV RNA levels were measured using the Roche COBAS® AmpliPrep/COBAS® TaqMan® HCV Test, v2.0 assay, which has a LLoQ of 15 IU/mL.
Time Frame: Up to 40 weeks
Population: All randomized participants who received at least 1 dose of study drug and had SVR24 results available are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | A1: GT1 NC GZR+UPR+EBR (8 Weeks) | A2: GT1 NC GZR+UPR+RZR (8 Weeks) | A3: GT2 NC GZR+UPR+EBR (8 Weeks) | A4: GT2 NC GZR+UPR+RZR (8 Weeks) | A5: GT1 NC GZR+UPR+EBR (8 Weeks) | A6: GT1 NC GZR+UPR+RZR (8 Weeks) | B6: GT1 NC GZR+UPR+RVR (8 Weeks) | A7: GT2 NC GZR+UPR+EBR (8 Weeks) | A8: GT2 NC GZR+UPR+RZR (8 Weeks) | B8: GT2 NC GZR+UPR+RZR (8 Weeks) | B9: GT1 NC GZR+UPR+RZR (12 Weeks) | B10: GT2 NC GZR+UPR+RZR (8 Weeks) + RBV | B11: GT2 NC GZR+UPR+RZR (12 Weeks) | B12: GT1 C GZR+UPR+RZR (8 Weeks) | B13: GT1 C GZR+UPR+RZR (12 Weeks) | B14: GT2 C GZR+UPR+RZR (12 Weeks) | B15: GT2 C GZR+UPR+RZR (12 Weeks) + RBV | 16: GT2 C GZR+UPR+RZR (16 Weeks)
Number analyzed (Participants) | 23 | 24 | 16 | 14 | 23 | 22 | 30 | 15 | 16 | 16 | 48 | 30 | 29 | 35 | 35 | 15 | 16 | 25
Percentage of Participants | 100.0 [85.2 to 100.0] | 100.0 [85.8 to 100.0] | 68.8 [41.3 to 89.0] | 71.4 [41.9 to 91.6] | 100.0 [85.2 to 100.0] | 90.9 [70.8 to 98.9] | 100.0 [88.4 to 100.0] | 60.0 [32.3 to 83.7] | 93.8 [69.8 to 99.8] | 87.5 [61.7 to 98.4] | 100.0 [92.6 to 100.0] | 83.3 [65.3 to 94.4] | 100.0 [88.1 to 100.0] | 97.1 [85.1 to 99.9] | 100.0 [90.1 to 100.0] | 100.0 [78.2 to 100.0] | 100.0 [79.4 to 100.0] | 100.0 [86.3 to 100.0]

4. Primary Outcome: Percentage of Participants Discontinuing From Study Treatment Due to an AE
Description: as for outcome 2
Time Frame: Up to 16 weeks
Population: All randomized participants who received at least 1 dose of study drug are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | A1: GT1 NC GZR+UPR+EBR (8 Weeks) | A2: GT1 NC GZR+UPR+RZR (8 Weeks) | A3: GT2 NC GZR+UPR+EBR (8 Weeks) | A4: GT2 NC GZR+UPR+RZR (8 Weeks) | A5: GT1 NC GZR+UPR+EBR (8 Weeks) | A6: GT1 NC GZR+UPR+RZR (8 Weeks) | B6: GT1 NC GZR+UPR+RVR (8 Weeks) | A7: GT2 NC GZR+UPR+EBR (8 Weeks) | A8: GT2 NC GZR+UPR+RZR (8 Weeks) | B8: GT2 NC GZR+UPR+RZR (8 Weeks) | B9: GT1 NC GZR+UPR+RZR (12 Weeks) | B10: GT2 NC GZR+UPR+RZR (8 Weeks) + RBV | B11: GT2 NC GZR+UPR+RZR (12 Weeks) | B12: GT1 C GZR+UPR+RZR (8 Weeks) | B13: GT1 C GZR+UPR+RZR (12 Weeks) | B14: GT2 C GZR+UPR+RZR (12 Weeks) | B15: GT2 C GZR+UPR+RZR (12 Weeks) + RBV | 16: GT2 C GZR+UPR+RZR (16 Weeks)
Number analyzed (Participants) | 23 | 24 | 16 | 14 | 23 | 23 | 30 | 15 | 16 | 16 | 48 | 31 | 31 | 35 | 40 | 15 | 16 | 26
Percentage of Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6.5 | 0 | 0 | 2.5 | 0 | 12.5 | 0

ADVERSE EVENTS:
Time Frame: Up to 18 weeks (14 days after completing treatment)
Description: All participants who received at least 1 dose of study drug are included.
Groups:
- B10: GT2 NC GZR+UPR+RZR (8 Weeks) + RBVMax 62 Characters...: In Part B, HCV GT2-infected NC participants took 2 FDC tablets containing GZR 50 mg + UPR 225 mg + RZR 30 mg per tablet q.d. by mouth for 8 weeks. Participants will also take RBV b.i.d. at a total daily dose of 800-1600 mg based on body weight.
Arm/Group | A1: GT1 NC GZR+UPR+EBR (8 Weeks) | A2: GT1 NC GZR+UPR+RZR (8 Weeks) | A3: GT2 NC GZR+UPR+EBR (8 Weeks) | A4: GT2 NC GZR+UPR+RZR (8 Weeks) | A5: GT1 NC GZR+UPR+EBR (8 Weeks) | A6: GT1 NC GZR+UPR+RZR (8 Weeks) | A7: GT2 NC GZR+UPR+EBR (8 Weeks) | A8: GT2 NC GZR+UPR+RZR (8 Weeks) | B6: GT1 NC GZR+UPR+RVR (8 Weeks) | B8: GT2 NC GZR+UPR+RZR (8 Weeks) | B9: GT1 NC GZR+UPR+RZR (12 Weeks) | B10: GT2 NC GZR+UPR+RZR (8 Weeks) + RBVMax 62 Characters... | B11: GT2 NC GZR+UPR+RZR (12 Weeks) | B12: GT1 C GZR+UPR+RZR (8 Weeks) | B13: GT1 C GZR+UPR+RZR (12 Weeks) | B14: GT2 C GZR+UPR+RZR (12 Weeks) | B15: GT2 C GZR+UPR+RZR (12 Weeks) + RBV | B16: GT2 C GZR+UPR+RZR (16 Weeks)
Serious Adverse Events (participants affected / at risk) | 0/23 | 1/24 | 1/16 | 1/14 | 0/23 | 0/23 | 0/15 | 0/16 | 0/30 | 1/16 | 0/48 | 2/31 | 0/31 | 1/35 | 3/40 | 0/15 | 0/16 | 2/26
Other Adverse Events (participants affected / at risk) | 13/23 | 19/24 | 10/16 | 10/14 | 15/23 | 13/23 | 13/15 | 12/16 | 18/30 | 11/16 | 35/48 | 24/31 | 19/31 | 19/35 | 26/40 | 8/15 | 13/16 | 14/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A1: GT1 NC GZR+UPR+EBR (8 Weeks) (N=23) | A2: GT1 NC GZR+UPR+RZR (8 Weeks) (N=24) | A3: GT2 NC GZR+UPR+EBR (8 Weeks) (N=16) | A4: GT2 NC GZR+UPR+RZR (8 Weeks) (N=14) | A5: GT1 NC GZR+UPR+EBR (8 Weeks) (N=23) | A6: GT1 NC GZR+UPR+RZR (8 Weeks) (N=23) | A7: GT2 NC GZR+UPR+EBR (8 Weeks) (N=15) | A8: GT2 NC GZR+UPR+RZR (8 Weeks) (N=16) | B6: GT1 NC GZR+UPR+RVR (8 Weeks) (N=30) | B8: GT2 NC GZR+UPR+RZR (8 Weeks) (N=16) | B9: GT1 NC GZR+UPR+RZR (12 Weeks) (N=48) | B10: GT2 NC GZR+UPR+RZR (8 Weeks) + RBVMax 62 Characters... (N=31) | B11: GT2 NC GZR+UPR+RZR (12 Weeks) (N=31) | B12: GT1 C GZR+UPR+RZR (8 Weeks) (N=35) | B13: GT1 C GZR+UPR+RZR (12 Weeks) (N=40) | B14: GT2 C GZR+UPR+RZR (12 Weeks) (N=15) | B15: GT2 C GZR+UPR+RZR (12 Weeks) + RBV (N=16) | B16: GT2 C GZR+UPR+RZR (16 Weeks) (N=26)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal artery occlusion (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pilonidal cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Substance-induced psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A1: GT1 NC GZR+UPR+EBR (8 Weeks) (N=23) | A2: GT1 NC GZR+UPR+RZR (8 Weeks) (N=24) | A3: GT2 NC GZR+UPR+EBR (8 Weeks) (N=16) | A4: GT2 NC GZR+UPR+RZR (8 Weeks) (N=14) | A5: GT1 NC GZR+UPR+EBR (8 Weeks) (N=23) | A6: GT1 NC GZR+UPR+RZR (8 Weeks) (N=23) | A7: GT2 NC GZR+UPR+EBR (8 Weeks) (N=15) | A8: GT2 NC GZR+UPR+RZR (8 Weeks) (N=16) | B6: GT1 NC GZR+UPR+RVR (8 Weeks) (N=30) | B8: GT2 NC GZR+UPR+RZR (8 Weeks) (N=16) | B9: GT1 NC GZR+UPR+RZR (12 Weeks) (N=48) | B10: GT2 NC GZR+UPR+RZR (8 Weeks) + RBVMax 62 Characters... (N=31) | B11: GT2 NC GZR+UPR+RZR (12 Weeks) (N=31) | B12: GT1 C GZR+UPR+RZR (8 Weeks) (N=35) | B13: GT1 C GZR+UPR+RZR (12 Weeks) (N=40) | B14: GT2 C GZR+UPR+RZR (12 Weeks) (N=15) | B15: GT2 C GZR+UPR+RZR (12 Weeks) + RBV (N=16) | B16: GT2 C GZR+UPR+RZR (16 Weeks) (N=26)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Excessive cerumen production (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Androgen deficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharospasm (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 5 (5) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1) | 2 (3) | 3 (3) | 0 (0) | 6 (8) | 3 (3) | 5 (5) | 2 (3) | 7 (7) | 5 (6) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 3 (3) | 4 (4)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (3)
Asthenia (General disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (5) | 1 (2)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Crying (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Drug withdrawal syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Energy increased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (5) | 3 (3) | 2 (2) | 2 (2) | 6 (6) | 4 (4) | 6 (6) | 6 (6) | 4 (4) | 3 (4) | 8 (9) | 4 (4) | 1 (1) | 3 (3) | 3 (3) | 1 (1) | 5 (5) | 3 (4)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 1 (2)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sialoadenitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulse abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 3 (3) | 1 (2) | 3 (3) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 2 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (5) | 7 (9) | 3 (4) | 2 (2) | 8 (9) | 3 (4) | 5 (5) | 9 (10) | 2 (2) | 3 (3) | 15 (25) | 8 (8) | 7 (7) | 5 (6) | 5 (11) | 2 (2) | 2 (2) | 4 (10)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Affective disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Flat affect (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Initial insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (3) | 2 (2) | 3 (3) | 1 (1) | 4 (5) | 4 (4) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 1 (1)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mood altered (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Menstruation delayed (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart rate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Essential hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation.